CLINICAL TRIAL: NCT00004239
Title: A Phase I Study of Compound 506U78 (NSC #686673) in Patients With Hematologic Malignancies and Renal or Hepatic Impairment
Brief Title: 506U78 in Treating Patients With Hematologic Cancer and Kidney or Liver Impairment
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: poor accrual
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-69803; U10CA031946 (NIH); CLB-69803; CDR0000067483 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2000-01-28; First posted 2004-01-29 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: recurrent adult Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; refractory multiple myeloma; Waldenstrom macroglobulinemia; stage III multiple myeloma; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; polycythemia vera; primary myelofibrosis; essential thrombocythemia; refractory hairy cell leukemia; chronic myelomonocytic leukemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult T-cell leukemia/lymphoma; previously treated myelodysplastic syndromes; prolymphocytic leukemia; primary systemic amyloidosis; recurrent mantle cell lymphoma; anaplastic large cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Waldenstrom Macroglobulinemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Leukemia, Hairy Cell; Leukemia, Myelomonocytic, Chronic; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Immunoglobulin Light-chain Amyloidosis; Lymphoma, Mantle-Cell; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone | interventions — nelarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Compound 506U78 (Experimental): Compound 506U78 will be administered intravenously over 2 hours on days 1, 3 and 5 of each 28 day treatment cycle.
  Interventions: Drug: Compound 506U78

INTERVENTIONS:
Drug: Compound 506U78

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of 506U78 in treating patients who have hematologic cancer and kidney or liver impairment.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of 506U78 in patients with hematologic malignancies and renal or hepatic impairment. II. Establish dosing guidelines for this drug in this patient population. III. Determine the toxicities and pharmacokinetics of this drug in these patients.

OUTLINE: Patients are stratified into 5 groups according to renal and hepatic function: Group 1: Normal renal function and normal hepatic function Group 2: Moderate renal impairment and normal hepatic function Group 3: Severe renal impairment and normal hepatic function Group 4: End stage renal impairment and normal hepatic function Group 5: Normal renal function and moderate hepatic impairment Group 1: Patients receive 506U78 IV over 2 hours on days 1, 3, and 5. Groups 2-5: Patients receive 506U78 IV over 2 hours on days 1, 3, and 5. Dose escalation occurs independently in each of the treatment groups. Cohorts of 3-6 patients receive escalating doses of 506U78 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicities. Treatment repeats every 4 weeks for a maximum of 6 courses in the absence of unacceptable toxicity or disease progression.

PROJECTED ACCRUAL: Approximately 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed hematologic malignancy that has failed standard therapy or for which no standard therapy exists, including, but not limited to, the following: Acute lymphocytic leukemia Acute myelogenous leukemia Chronic lymphocytic leukemia Chronic myelogenous leukemia Multiple myeloma Non-Hodgkin's lymphoma Hodgkin's disease No history of CNS disease, including carcinomatous meningitis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: CTC 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin: Groups 1-4: Less than 1.5 times upper limit of normal (ULN) Group 5: 1.5-4 times ULN Renal: Creatinine clearance: Groups 1 and 5: Greater than 50 mL/min Group 2: 30-50 mL/min Group 3: Less than 30 mL/min Group 4: Less than 30 mL/min, requiring dialysis Neurologic: No history of grade 2 peripheral neuropathy No history of seizure disorder No history of neurologic dysfunction Other: Not pregnant or nursing Fertile patients must use effective contraception HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy (e.g., interferon, monoclonal antibodies) No concurrent interleukin-11 for treatment or prevention of thrombocytopenia No concurrent prophylactic colony stimulating factors Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks for melphalan, carmustine, or mitomycin) At least 72 hours since prior hydroxyurea No prior 506U78 No other concurrent chemotherapy Endocrine therapy: At least 72 hours since prior glucocorticoids Concurrent continuation of steroids for adrenal failure allowed No concurrent hormones except for nondisease related conditions (e.g., insulin for diabetes) No concurrent dexamethasone or other steroidal antiemetics Radiotherapy: At least 4 weeks since prior radiotherapy No concurrent palliative radiotherapy No concurrent whole brain irradiation for documented CNS disease Surgery: Not specified Other: At least 72 hours since prior aspirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 1999-12; Primary Completion 2002-01 (Actual); Study Completion 2002-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Todd M. Zimmerman, MD, Study Chair — University of Chicago
Locations (3):
- United States (3):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina